CLINICAL TRIAL: NCT06024421
Title: EVALUATION DE LA TOLERANCE ET DU PROFIL PHARMACOCINETIQUE DE DOSES ELEVEES DE FAVIPIRAVIR CHEZ LE VOLONTAIRE SAIN
Brief Title: Evaluation of Tolerance and Pharmacokinetic Profile of High Doses of Favipiravir in Healthy Volunteers
Acronym: FAVIDOSE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: FUJIFILM Toyama Chemical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C18-47; 2022-502871-49-00 (Other: EU CT)
Record Dates: First submitted 2023-07-07; First posted 2023-09-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Infectious Disease; Pharmacology
Keywords: healthy volunteer; dose escalation; tolerance; pharmacokinetics; favipiravir
MeSH Terms: conditions — Communicable Diseases | interventions — favipiravir

STUDY DESIGN:
Intervention Model Description: Dose-escalation trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active and placebo will not be visually distinguishable. Packaging and labeling of active and placebo tablets will be done in such a way as to not allow unblinding without access to the randomization list or the investigational drug unit list.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- level 1: experimental (Experimental): D1: 2400 mg BID; D2 to D13: 1600 mg BID and D14: 1600 mg in the morning
  Interventions: Drug: favipiravir
- level 2: experimental (Experimental): D1: 2400 mg BID; D2 to D13: 2000 mg BID and D14: 2000 mg in the morning
  Interventions: Drug: favipiravir
- level 3: experimental (Experimental): D1: 2400 mg BID; D2 to D13: 2400 mg BID andD14: 2400 mg in the morning
  Interventions: Drug: favipiravir
- level 1: placebo (Placebo Comparator): D1: 2400 mg BID; D2 to D13: 1600 mg BID and D14: 1600 mg in the morning
  Interventions: Drug: Placebo
- level 2: placebo (Placebo Comparator): D1: 2400 mg BID; D2 to D13: 2000 mg BID and D14: 2000 mg in the morning
  Interventions: Drug: Placebo
- level 3: placebo (Placebo Comparator): D1: 2400 mg BID; D2 to D13: 2400 mg BID andD14: 2400 mg in the morning
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: favipiravir — Light yellow, film-coated tablet, each containing 200 mg of favipiravir
  Arms: level 1: experimental; level 2: experimental; level 3: experimental
Drug: Placebo — Light yellow, film-coated tablet
  Arms: level 1: placebo; level 2: placebo; level 3: placebo

SUMMARY:
FAVIDOSE trial is a Phase I randomized, double blind controlled, monocentric, dose escalation clinical trial. The primary purpose of this trial is to evaluate tolerance of high doses of favipiravir for 14 days in healthy volunteers. This trial also looks to characterize favipiravir pharmacokinetics in blood and favipiravir levels in sperm. A pharmacogenetics analysis will be conducted in an attempt to identify genetic variants of metabolism and transport enzymes of favipiravir to explain the inter-individual variability of pharmacokinetic parameters of favipiravir.

Three sequential dose levels including distinctive participants:

* level 1: D1: 2400 mg BID; D2 to D13: 1600 mg BID and D14: 1600 mg in the morning;
* level 2: D1: 2400 mg BID; D2 to D13: 2000 mg BID and D14: 2000 mg in the morning;
* level 3: D1: 2400 mg BID; D2 to D13: 2400 mg BID andD14: 2400 mg in the morning.

Three study groups of maximum of 8 participants, 6 receiving favipiravir and 2 receiving placebo per dose level, three dose levels proposed. Seven additional participants with the same follow up will be included and randomized (6:1 ratio) at the maximum tolerated dose level to allow a satisfactory accurate characterization of pharmacokinetics and pharmacogenetics of favipiravir and their determinants (maximum 39 participants in total, taking into account 8 participants - 2 per dose level - replaced because loss of follow-up before the end of treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Man between 50 and 75 years old without any desire to have children or woman between 18 and 75 years old ;
2. Subject considered healthy after a thorough general examination (questioning, physical examination);
3. For men: acceptance of semen collection by masturbation;
4. For men: acceptance of condom use from initiation of the investigational drug until 1 month after stopping the investigational drug;
5. For women of childbearing potential: effective contraceptive method combining two methods of contraception (one female contraceptive method combined with male condom use) from the inclusion visit until 1 month after discontinuation of the investigational drug;
6. Blood chemistry:

   * Kalemia, Calcemia, Prothrombin rate (PT), Activated partial thromboplastin time (APTT): values within laboratory normal;
   * ALT, ASAT, Uricemia: values below the upper limit of the laboratory normal;
   * Other biological results (Blood count; Natremia; Phosphoremia; Chloremia; Fasting blood glucose; Gamma glutamyl transpeptidase; Urea; Total bilirubin; Creatinine; CPK; Lactate dehydrogenase; Albuminemia; Proteinemia; Triglycerides; C-reactive protein; Albumin/Globulin ratio; Alkaline phosphatase) with no clinically significant abnormality.

   NB: A parameter outside the usual values considered clinically significant may, at the investigator's discretion, be tested a second time on another sample taken outside of a visit planned in the protocol before the initiation of the experimental drug.
7. Urine dipstick (biochemistry: leukocyturia, proteinuria and hematuria) without clinically significant abnormality;
8. Urine tox screen negative (amphetamines/metamphetamines, barbiturates, benzodiazepines, cannabis, cocaine, opiates);
9. Ability to take the investigational drug orally and adherence to the dosage of the investigational drug;
10. Acceptance and signing of the informed consent;
11. Membership in a social security plan or beneficiary of such a plan;
12. Adherence to lifestyle considerations (see section 5.5) during participation in this research.

Exclusion Criteria:

1. Concomitant use or within 15 days prior to inclusion of another QT/QTc prolonging drug or drugs that may disrupt electrolyte levels, among others: loop diuretics, thiazide diuretics and related drugs (see list www.crediblemeds.org)
2. History of amiodarone use within 6 months prior to inclusion
3. History of gout or current treatment for gout or hyperuricemia
4. Treatment with pyrazinamide or any other drug known to induce hyperuricemia
5. History of hypersensitivity reaction to a nucleoside analog targeting viral RNA polymerase
6. Known hypersensitivity to any of the components (favipiravir or placebo)
7. Pregnant or breastfeeding women
8. For men: history of vasectomy or known history of infertility.
9. Refusal of the subject to complete all the visits, clinical and paraclinical examinations planned by the study
10. On ECG: PR >200ms, QRS >100ms QTc >450ms and morphological appearance of abnormal repolarization
11. PAS <100 mmHg
12. Any history or active cardiovascular, pulmonary, intestinal, hepatic, renal, metabolic, hematologic, neurologic, bone, joint, muscular, psychiatric, systemic, ocular, gynecologic, andrologic, or infectious disease (including active HIV, HCV, or HBV infection), or any acute condition, which in the judgment of the investigator could be detrimental to the volunteer and/or interfere with or limit the protocol evaluation and data analysis
13. Personal or family history of long QT syndrome, torsades de pointes or sudden death
14. Patient with severe hepatic impairment
15. Gastrointestinal pathology such as ileus, colitis or enterocolitis
16. Treatment with another investigational drug or other investigational procedure (clinical trial, clinical investigation of a medical device, category 1 or 2 research involving humans);
17. A person who is subject to a legal protection measure (safeguard of justice, curatorship, guardianship);
18. Person placed in administrative detention;
19. Person who, in the judgment of the investigating physician, may be non-observant during the study, or unable to communicate due to a language barrier or mental disorder
20. Person who cannot be contacted in an emergency
21. Person with at least one first-degree relative from East Asia or Southeast Asia.

Secondary Exclusion Criteria

Participants with at least one of the following criteria will not start the experimental treatment at D1 if they are already randomized:

1. Positive nasopharyngeal antigen test for SARS-CoV-2 at D1 (prior to treatment initiation)
2. Blood potassium levels outside the normal laboratory range within 8 days prior to treatment initiation (D1)
3. ECG: PR >200ms, QRS >100ms QTc >450ms and morphological appearance of abnormal repolarization on Day 1
4. Positive pregnancy test on Day 1 (before initiation of treatment)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Tolerance | Months 6
  Tolerance of high doses of favipiravir, defined by the number of participants with at least one adverse medical event considered as related to favipiravir (AER)-as determined and validated by the sponsor- clinical stage 3 or 4 according to the CTCAE (v5.0) not found at inclusion at same level and biological AER de stage 3 or 4 not found at inclusion in the same level. AER are collected daily until D15 and at D21 and D28, as well as at M3 and M6 for participating men.
  D1 is the first day of favipiravir or placebo intake.

SECONDARY OUTCOMES:
Plasma concentration of favipiravir | Day 1 (Hour 0; Hour 0.5 ; Hour 1; Hour 2; Hour 5; Hour 8), Day 3 (Hour 0 ; Hour 0.5; Hour 2), Day 7 (Hour 0; Hour 0.5 ; Hour 1; Hour 2; Hour 5; Hour 8), Day 10 (Hour 0), Day 14 (Hour 0; Hour 0.5 ; Hour 1; Hour 2; Hour 5; Hour 8), Day 15 (Hour 0)
  Construction of the pharmacokinetic model and the estimation of its parameters will be realized by a population pharmacokinetic analysis integrating all available data on plasma concentration.
Genetic | Days 1
  Genetic variants associated with favipiravir exposure. Targeted genotyping of variants of the gene encoding the enzyme responsible for transport and metabolism of favipiravir (aldehyde deshydrogenase) will be performed.
Sperm pharmacology | Day 14, day 28
  For participating men: favipiravir concentration in sperm at D14 and D28.

CONTACTS AND LOCATIONS:
Overall Officials: Denis MALVY, Study Chair — CHU de Bordeaux & INSERM, Université de Bordeaux, France; Xavier DUVAL, Principal Investigator — APHP Hôpital Bichat Claude Bernard; Jean-Jacques KILADJIAN, Study Director — INSERM Pôle Recherche Clinique
Locations (1):
- University Hospital Bichat - Claude Bernard, Paris, France